CLINICAL TRIAL: NCT05671549
Title: Evaluation of the Effects of Arthrocentesis Combined With Occlusal Stabilization Splint on Disc Displacement Without Reduction-induced Acute and Closed Lock. A Prospective Cohort Study
Brief Title: Combined Arthrocentesis and Occlusal Splint Therapy for Closed Locks of the TMJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Aras Erdil, Researcher in the related department, Tokat Gaziosmanpasa University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 83116987-381
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Arthrocentesis; Closed lock; Stabilization splint
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Closed-Lock (Active Comparator): The participants will be enrolled in this group regarding the duration (longer than three months) of their symptoms. The allocated participants will undergo one session of the arthrocentesis procedure. The prefabricated occlusal stabilization splints will be applied. The participants' preoperative, postoperative immediate, and postoperative seventh-day pain intensities and maximum mouth-opening amounts will be recorded and analyzed.
  Interventions: Procedure: Arthrocentesis of the temporomandibular joint
- Acute Closed-Lock (Active Comparator): The participants will be enrolled in this group regarding the duration (shorter than three months) of their symptoms. The allocated participants will undergo one session of the arthrocentesis procedure. The prefabricated occlusal stabilization splints will be applied. The participants' preoperative, postoperative immediate, and postoperative seventh-day pain intensities and maximum mouth-opening amounts will be recorded and analyzed.
  Interventions: Procedure: Arthrocentesis of the temporomandibular joint

INTERVENTIONS:
Procedure: Arthrocentesis of the temporomandibular joint — Arthrocentesis of the temporomandibular joint is a minimally invasive method performed under local anesthesia to irrigate the upper temporomandibular joint cavity with biocompatible substances. The procedure aims to wash out intra-articular inflammatory substances, reduce pain and restore the function of the related joint.

SUMMARY:
The goal of this prospective cohort study is to evaluate the effectiveness of combined arthrocentesis and occlusal stabilization splint therapy in patients diagnosed with disc displacement without reduction of temporomandibular joint-induced closed locks. The main questions it aims to answer are:

* Is there a difference in the treatment response between chronic and acute closed-lock conditions?
* On which dimensions of pain did the treatment have positive effects? Participants will be preoperatively examined and assigned to one of the two study groups.
* All participants undergo a single session of TMJ arthrocentesis.
* Following the arthrocentesis session, all participants will use preoperatively fabricated occlusal splints.
* Participants will be recalled in one week to evaluate the outcomes. Researchers will compare acute and chronic closed-lock groups to see if there are differences between pain intensities and mouth-opening amounts postoperatively.

DETAILED DESCRIPTION:
The study sample constituted patients diagnosed with DDWoR with limited opening according to the Turkish version of the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD Axis 1 questionnaire and examination form). The included patients with DDWoR-induced complaints persisting for more than three months were considered chronic (Group 1), and those with a shorter duration were considered acute (Group 2). For clinical diagnosis of DDWoR, Significant limitation of mouth opening, less than 35 mm assisted mouth opening, less than 4 mm increase in mouth opening with passive stretching, less than 7 mm contralateral movement of the mandible, and deviation of the mandible to the affected side during mouth opening was considered sufficient. The DC/TMD questionnaire and clinical examination diagnoses were confirmed by magnetic resonance images (MRI).

Preoperative and postoperative clinical examinations consisted of recording demographic information, amount of maximum mouth opening (MMO), and determination of McGill Pain Questionnaire (MPQ) and Visual Analog Scale (VAS) scores. MMO values were determined as the distance between the incisal edges of upper and lower central teeth and recorded in millimeters. MPQ scores were obtained with the questionnaire form consisting of four subsections. In the first subsection of the questionnaire, besides the patient's demographic data, the location of the current pain and whether it comes from superficial or deep tissues are questioned. In the second subsection, there are 20-word groups containing 78 words that ask the Sensory (groups 1-10), Affective (groups 11-15), Evaluative (group 16), and Miscellaneous (groups 17-20) components of current pain. In the third subsection, the relationship of pain with time is questioned. There are word groups to determine the continuity of pain, its frequency, and factors that increase or reduce pain. In the fourth subsection, five-word groups ranging from "mild" pain to "unbearable" pain to determine the severity of the pain; There are also six questions to assess the severity of pain that the patient can accept or experience without discomfort, which is also defined as "experienceable=target pain." The obtainable MPQ scores range from 0 to 78. The higher the scores, the greater the pain. Also, preoperative and postoperative VAS scores were obtained by marking a point on a 10 cm line. The score was calculated as the distance in centimeters between the zero and the marked points.

ELIGIBILITY:
Inclusion Criteria:

* individuals over the age of 18
* completion of the arthrocentesis treatment without any complications;
* the presence of preoperative information and postoperative follow-up data;
* persistent complaints despite conservative methods (behavioral modification, diet restrictions, non-steroid anti-inflammatory drugs, and physical therapy) for at least three months.

Exclusion Criteria: The patients;

* diagnosed with any connective tissue, neurological, dermatological, inflammatory diseases, and TMD other than DDWoR,
* who underwent TMJ surgeries, arthrocentesis procedures, TMJ ankylosis surgery,
* previously used occlusal splints,
* who developed complications in the application of arthrocentesis in the current study (low-volume lavage, extravasation, inability to reach the upper joint space, e.g.),
* with lack of teeth to affect the fabrication of the occlusal stabilization splint,
* with a history of radiotherapy of the head and neck.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Baseline Pain intensity with Visual analog scale | At the initial visit before arthrocentesis procedure.
  The pain intensity measurement was performed with the Visual analog scale (VAS), in which 0 referred to 'no pain,' 5 referred to 'moderate pain,' and ten referred to 'excruciating pain.' The patients were asked to mark their pain intensities on the VAS scale.
Baseline Pain intensity with McGill pain questionnaire | At the initial visit before arthrocentesis procedure.
  The pain intensity measurement was performed with the McGill Pain Questionnaire form. According to the word groups chosen by the participants, the total score of the questionnaire varies between 0-78. An increase in the total score is interpreted as the severity of pain intensity.
Change From Baseline Maximum Mouth Opening on Postoperative Follow Up Visits | At the initial visit, at the session of arthrocentesis postoperatively, at the first week
  All patients' maximal mouth opening were measured and recorded as the distance between upper and lower right central incisors.
Postoperative Pain intensity with Visual analog scale | At first week follow-up visit
  The pain intensity measurement was performed with the Visual analog scale (VAS), in which 0 referred to 'no pain,' 5 referred to 'moderate pain,' and ten referred to 'excruciating pain.' The patients were asked to mark their pain intensities on the VAS scale.
Postoperative Pain intensity with McGill pain questionnaire | At first week follow-up visit
  The pain intensity measurements were performed with the McGill Pain Questionnaire form. According to the word groups chosen by the participants, the total score of the questionnaire varies between 0-78. An increase in the total score is interpreted as the severity of pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet K. Tümer, AssocProfDr, Study Director — Alanya Alaaddin Keykubat University
Locations (1):
- Tokat Gaziosmanpasa University, Faculty of Dentistry, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data regarding participants were made available in the manuscript

REFERENCES:
- [Background] Hosgor H. Is arthrocentesis plus hyaluronic acid superior to arthrocentesis alone in the treatment of disc displacement without reduction in patients with bruxism? J Craniomaxillofac Surg. 2020 Nov;48(11):1023-1027. doi: 10.1016/j.jcms.2020.07.008. Epub 2020 Jul 25. PMID 33028488
- [Result] Tatli U, Benlidayi ME, Ekren O, Salimov F. Comparison of the effectiveness of three different treatment methods for temporomandibular joint disc displacement without reduction. Int J Oral Maxillofac Surg. 2017 May;46(5):603-609. doi: 10.1016/j.ijom.2017.01.018. Epub 2017 Feb 20. PMID 28222947
- [Derived] Erdil A, Demirsoy MS, Tumer MK. Evaluation of the effects of arthrocentesis combined with occlusal stabilization splint on disc displacement without reduction-induced acute and closed lock. A prospective cohort study. J Stomatol Oral Maxillofac Surg. 2023 Oct;124(5):101438. doi: 10.1016/j.jormas.2023.101438. Epub 2023 Mar 12. PMID 36918123